CLINICAL TRIAL: NCT05243771
Title: Norwegian Stoma Trial - Open-label, Multicenter Trial
Brief Title: Norwegian Stoma Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of North Norway (Other); Helse Nord-Trøndelag HF (Other); St. Olavs Hospital (Other); Alesund Hospital (Other); Helse Fonna (Other); Helse Stavanger HF (Other Government); Sorlandet Hospital HF (Other Government); Sykehuset Telemark (Other Government); Vestre Viken Hospital Trust (Other); Asker & Baerum Hospital (Other); Ullevaal University Hospital (Other); Oslo University Hospital (Other); Ostfold Hospital Trust (Other); University Hospital, Akershus (Other); Hamar Hospital (Unknown); Gjøvik Hospital (Unknown); Bodø Hospital (Unknown)
Responsible Party: Principal Investigator, Lars Thomas, Principal Investigator, The Hospital of Vestfold
Other Study IDs: 21/05179
Record Dates: First submitted 2022-01-11; First posted 2022-02-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer; Ileostomy; Complications; Quality of Life; Complication,Postoperative
MeSH Terms: conditions — Rectal Neoplasms; Postoperative Complications | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rectal resection with diverting stoma: Patients operated for rectal cancer with rectal resection and diverting stoma.
  Interventions: Procedure: Rectal resection with diverting stoma
- Rectal resection without diverting stoma: Patients operated for rectal cancer with rectal resection without diverting stoma.
  Interventions: Procedure: Rectal resection without diverting stoma
- Rectal resection with primary colostomy: Patients operated for rectal cancer with rectal resection with primary colostomy.
  Interventions: Procedure: Rectal resection with permanent colostomy

INTERVENTIONS:
Procedure: Rectal resection with diverting stoma — Patients in this group will receive a rectal resection with an anastomosis and also a diverting stoma will be created
  Groups: Rectal resection with diverting stoma
Procedure: Rectal resection without diverting stoma — Patients in this group will receive a rectal resection with an anastomosis and no diverting stoma will be created
  Groups: Rectal resection without diverting stoma
Procedure: Rectal resection with permanent colostomy — Patients in this group will receive a rectal resection and a permanent colostomy will be created
  Groups: Rectal resection with primary colostomy

SUMMARY:
The Norwegian Stoma Trial is an open-label multicenter trial investigating the use of stomas, both diveriting and permanent, in the surgical treatment of rectal cancer. The objective is to compare the chosen strategy to surgical complications, health realted quality of life and length of stay.

DETAILED DESCRIPTION:
In this national, multicenter study the study group will investigate whether patients with rectal adenocarcinoma undergoing a resection with an anastomosis will benefit from a diverting stoma or not, by studying how choice of surgery affects complications. In addition the study group will investigate complication rates and HRQoL among patients receiving a permanent colostomy and compare this to patients who have received an anastomosis. The investigators know that there are different approaches to the use of stomas (both permanent and diverting) between different hospitals. The investigators aim to discover potential differences in complication rates, length of stay and HRQoL among these patients and compare this to the chosen strategy. Health related quality of life will be measured using the EORTC CR 29 and EORTC CR 30 questionnares. Bowel function will also be monitored using the LARS (low anterior resection syndrome) score.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Verified rectal adenocarcinoma by biopsy
* Tumor located in the rectum with lower border of the tumor located 15 cm or less from the anal verge.
* Given informed consent

Exclusion Criteria:

* Advanced tumor stage requiring exenterative surgery beyond a convetional APR or TME.
* Stage IV disease
* Synchronous colon cancer necessitating a total colectomy
* Other concomitant disease(s) which will complicate participation.
* Unwillingness to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing a formal resection for rectal cancer will be asked to participate as long as they fit the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Surgical complications graded as Accordion grade 3 or more | Measured one year after the primary surgery
  The study group will investigate whether patients undergoing rectal resection with an anastomosis with a diverting stoma will have higher complication rates compared to patients who do not recieve a diverting stoma.

SECONDARY OUTCOMES:
Total length of hospital stay | Measured one year after the primary surgery
  Number of days admitted at hospital. The study group will investigate whether patients undergoing rectal resection with an anastomosis with a diverting stoma will have a higher number of days admitted to hospital compared to patients who do not recieve a diverting stoma.
Generic health related quality of life measured by the European Organization for Research and Treatment of Cancer (EORTC) C30 questionnaire | One year after the primary surgery
  Generic health related quality of life is measured using the EORTC C30 questionnaire. Investigate whether patients receiving a rectal resection with a primary colostomy have poorer health related quality of life compared to patients receiving an anastomosis.
Bowel function measured by the Low Anterior Resection Syndrome (LARS) score | One year after the primary surgery
  Bowel function is measured using the Low Anterior Resection Syndrome score. The score ranges from 0 to 42 points The higher the score, the worse the bowel function. Investigate whether patients undergoing rectal resection with an anastomosis with a diverting stoma will have higher LARS scores compared to patients who do not recieve a diverting stoma.
Surgical complications graded as Accordion grade 3 or more | Measured one year after the primary surgery
  Investigate whether patients receiving a rectal resection with a primary colostomy have lower complication rates compared to patients receiving an anastomosis
Generic health related quality of life measured by the European Organization for Research and Treatment of Cancer (EORTC) C30 questionnaire. | One year after the primary surgery
  Generic health related quality of life is measured using the EORTC C30 questionnaire. Investigate whether patients undergoing rectal resection with an anastomosis with a diverting stoma will have poorer health related quality of life compared to patients who do not recieve a diverting stoma.
Disease specific health related quality of life measured by the European Organization for Research and Treatment of Cancer (EORTC) CR29 questionnnaire | One year after the primary surgery
  Disease specific health related quality of life measured by the EORTC CR29 questionnnaire. Investigate whether patients undergoing rectal resection with an anastomosis with a diverting stoma will have poorer health related quality of life compared to patients who do not recieve a diverting stoma.
Disease specific health related quality of life measured by the European Organization for Research and Treatment of Cancer (EORTC) CR29 questionnnaire. | One year after the primary surgery
  Disease specific health related quality of life measured by the EORTC CR29 questionnnaire. Investigate whether patients receiving a rectal resection with a primary colostomy have poorer health related quality of life compared to patients receiving an anastomosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Thomas Seeberg, MD, PhD, Principal Investigator — The Hospital of Vestfold
Locations (18):
- Norway (18):
  - Asker og Baerum Hospital, Bærums verk, Gjettum
  - Østfold Hospital Trust, Sarpsborg, Grålum
  - Akershus University Hospital, Oslo, Lørenskog
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Bodø Hospital, Bodø
  - Vestre Viken Hospital Trust, Drammen
  - Gjøvik Hospital, Gjøvik
  - Hamar Hospital, Hamar
  - Helse Fonna, Haugesund
  - Sorlandet Hospital HF, Kristiansand
  - Helse Nord-Trøndelag HF, Levanger
  - Ullevaal University Hospital, Oslo
  - Sykehuset Telemark, Skien
  - Helse Stavanger HF, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim
  - Vestfold Hospital Trust, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided